CLINICAL TRIAL: NCT04251481
Title: Assessment of the Role of Diffusion MRI Changes During Chemoradiation Treatment of Head and Neck Cancer
Brief Title: Diffusion MRI for Head and Neck Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-01454
Record Dates: First submitted 2020-01-08; First posted 2020-02-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Head Cancer Neck
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; Contrast Media; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimization of Techniques (Experimental): To optimize the diffusion MRI methods for assessment of cell viability, metabolism and perfusion in head and neck cancer. There will be 24 subjects enrolled for 2 year duration. Treatment-naïve patients with cervical metastatic lymph nodes (diameter > 10 mm) of HNSCC will be recruited to have one research PET/MR scan (including dMRI) and one dMRI-only scan within three days prior to treatment. These data will be used to optimize the dMRI method and assess the repeatability.
  Interventions: Radiation: PET/MRI with FDG; Radiation: MRI scan without contrast
- : Longitudinal Monitoring (Experimental): To assess the feasibility of using diffusion MRI metrics at early stages of treatment for prediction of treatment response in head and neck cancer patients undergoing standard-of-care chemoradiation therapy. There will be 36 subjects enrolled for 3 year duration. The study will do bi-weekly measurement to monitor tumor response longitudinally. This study will be restricted to treatment-naïve patients who present pathologically confirmed HNSCC with metastatic lymph nodes and who are scheduled to receive standard care of radiation therapy with concurrent chemotherapy. The patients enrolled in this arm of the study will have 4 dMRI scans. The imaging data for each patient will be the proposed dMRI measures at the baseline and their changes at each follow-up time period. DCE-MRI will be included in the baseline scan for tumor delination as in standard-of-care cancer imaging and to compare with the proposed dMRI method.
  Interventions: Radiation: MRI scan without contrast; Radiation: MRI with gadolinium

INTERVENTIONS:
Radiation: PET/MRI with FDG — For the PET/MRI scans, an intravenous (IV) catheter (thin tube) will be used to administer dyes (contrast) for both the MRI and PET portions of the examination. The dye for the PET portion will be 18F-fluorodeoxyglucose (FDG). FDG is an FDA-approved radioactive substance (isotope) that contains chemicals that can be traced by PET/MRI. The dye for the MRI portion will be a gadolinium based contrast medium which is also an FDA-approved substance that makes certain tissues, abnormalities or disease processes more clearly visible on MRI scans. MRI uses a strong magnetic field to create images of the body. Subjects will be asked to lie on a table that will slide into the scanner; Wear earplugs to reduce the noise made by the MRI scanner and lie still throughout the time in the scanner.
  Arms: Optimization of Techniques
Radiation: MRI scan without contrast — MRI uses a strong magnetic field to create images of the body. Subjects will be asked to lie on a table that will slide into the scanner to scan the neck ; Wear earplugs to reduce the noise made by the MRI scanner and lie still throughout the time in the scanner.
Radiation: MRI with gadolinium — For the MRI scans, an intravenous (IV) catheter (thin tube) will be used to administer dyes (contrast) for MR scans. The dye for the MRI will be a gadolinium based contrast medium which is also an FDA-approved substance that makes certain tissues, abnormalities or disease processes more clearly visible on MRI scans. MRI uses a strong magnetic field to create images of the body. Subjects will be asked to lie on a table that will slide into the scanner; Wear earplugs to reduce the noise made by the MRI scanner and lie still throughout the time in the scanner.
  Arms: : Longitudinal Monitoring

SUMMARY:
The proposed study is to investigate the feasibility of using quantitative diffusion MRI (dMRI) methods for accurate and comprehensive assessment of treatment response. dMRI is a powerful tool to probe treatment-induced change in tumors. It is a unique in vivo imaging technique sensitive to cellular microstructures at the scale of water diffusion length on the order of a few microns. Previous studies have shown that both diffusion coefficient D and diffusional kurtosis coefficient K are promising imaging markers of (i) cell viability which can be used for evaluation of early treatment response. However, it is often underappreciated that these dMRI metrics are not fixed constants, but rather functions of the diffusion time t, D(t) and K(t); their t-dependency is determined by tissue properties, such as cell size and membrane permeability of tissue. D(t) and K(t) of tumors can vary substantially depending on t in the range of diffusion times (30-100 ms) typically used in clinical scan.

DETAILED DESCRIPTION:
This study will investigate the t-dependency of dMRI over a range of diffusion times (30-500 ms) to determine an optimal diffusion time for treatment response assessment when only one diffusion time needs to be used, particularly in routine clinical studies. Furthermore, the data with multiple diffusion times will also be used to measure the water exchange time of cancer cells. Exchange time has been studied using Dynamic Contrast Enhanced (DCE) MRI by multiple groups including ours, and has been suggested as a marker of (ii) cellular metabolism that regulates the ATP-dependent ion channels co-transporting water molecules. The study will measure with dMRI, without using a contrast agent. The investigators also demonstrated that Intra-Voxel Incoherent Motion (IVIM) MRI metrics (pseudo diffusivity, Dp; perfusion fraction, fp), from multiple b-values at a fixed diffusion time, can be used to assess the perfusion status of tumor and they are also associated with tumor interstitial fluid pressure. The IVIM effect has been observed in various cancer types (33-39) and animal tumor models. The product fp*Dp - a quantity including both blood volume and velocity information - is considered as a parameter analogous to (iii) perfusion flow .

ELIGIBILITY:
Inclusion Criteria:

ARM 1

* Treatment-naïve HNSCC patients with metastatic lymph nodes prior to surgery or chemoradiation therapy
* Age 18 or older
* Subjects without capacity to consent will not be enrolled.
* Subjects will be asked to verbalize understanding of the key elements, for non-English speaking patients, institutional translation services will be utilized.

ARM 2

* Treatment-naïve HNSCC patients with metastatic lymph nodes who will undergo standard-of-care chemoradiation therapy
* Age 18 or older
* Subjects without capacity to consent will not be enrolled.
* Subjects will be asked to verbalize understanding of the key elements, for non-English speaking patients, institutional translation services will be utilized.

Exclusion Criteria:

* Subjects who have the following contraindications to MRI:
* Electrical implants such as cardiac pacemakers or perfusion pumps
* Ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial heart, valves with steel parts, metal fragments, shrapnel, bullets, tattoos near the eye, or steel implants
* History of seizures
* Patients with GFR < 15 ml/min/1.73m2 or who are on dialysis will be excluded from the study.
* Subjects who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Intra-class Correlation (ICC) | 6 weeks
  Estimated components from a random effects model in each dMRI measure will be used to compute intra-class correlation as estimates of repeatability of each measure.
Intra-subject Coefficient of Variation (CV) | 6 weeks
  Estimated components from a random effects model in each dMRI measure will be used to compute intra-subject coefficient of variation as estimates of repeatability of each measure.
Overall Response Rate (ORR) | 6 weeks
  Binary classification of treatment response as complete response (CR) versus partial response (PR) for participants at the end of the chemoradiation therapy assessed by clinical/radiological reports. CR will include the cases with complete disappearance of any clinically detectable tumor mass, while PR will include cases with stable disease and progressive disease.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 2 Years Post-Treatment
  Binary indicator of whether patients showed progression-free survival at 2 years post treatment on the standard-of-care follow-up exams. PFS is the length of time that a patient lives with the disease but it does not get worse.

CONTACTS AND LOCATIONS:
Overall Officials: Elcin Zan, MD, Principal Investigator — NYU Langone
Locations (2):
- United States (2):
  - NYU Langone, New York, New York
  - Weill Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to gene.kim@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.